CLINICAL TRIAL: NCT05168735
Title: Ketamine + Mindfulness for Depression
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rebecca Price (Other)
Responsible Party: Sponsor-Investigator, Rebecca Price, Associate Professor of Psychiatry and Psychology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY21110040
Record Dates: First submitted 2021-12-09; First posted 2021-12-23 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Depression, Unipolar
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous Ketamine + Mindfulness Exercises (Experimental)
  Interventions: Drug: Intravenous Ketamine; Behavioral: Brief Mindfulness Exercises
- Intravenous Ketamine + Academic Exercises (Active Comparator)
  Interventions: Drug: Intravenous Ketamine; Behavioral: Academic Exercises

INTERVENTIONS:
Drug: Intravenous Ketamine — Single infusion of intravenous racemic ketamine (0.5mg/kg over 40min)
Behavioral: Brief Mindfulness Exercises — 30min guided training in mindfulness meditation immediately prior to infusion
  Arms: Intravenous Ketamine + Mindfulness Exercises
Behavioral: Academic Exercises — 30min of mental math and other academic cognitive puzzles completed silently/mentally
  Arms: Intravenous Ketamine + Academic Exercises

SUMMARY:
In this project, the investigators will administer a single infusion of IV ketamine to depressed patients and randomize the patients to receive either a) usual/typical infusion conditions or b) mindfulness training and exercises in conjunction with the infusion. Investigators will test whether the conjunction of ketamine + mindfulness enhances the reductions in depression following a single ketamine infusion.

DETAILED DESCRIPTION:
NOTE: The study's target sample size was revised after beginning the study, based on a revised available budget.

ELIGIBILITY:
Inclusion Criteria:

All participants will:

1. be between the ages of 18 and 65 years,
2. score ≥ 14 on the Hamilton Depression Rating Scale (modified Ham-D)
3. possess a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign an informed consent document

Exclusion Criteria:

All participants:

1. Presence of lifetime bipolar, psychotic, or autism spectrum; current problematic substance use (e.g., ongoing moderate-to-severe substance use disorder);
2. Acute suicidality or other psychiatric crises requiring treatment escalation. We will use the Columbia Suicide Severity Rating Scale (CSSRS) as both an initial exclusion criteria (CSSRS "Baseline/Screening" Version for past 1month period) and as grounds for rescue/removal (CSSRS "Since Last Visit" form). The CSSRS will be administered using a paper form by an experienced and thoroughly trained clinical assessor on the study team. Subjects with CSSRS suicide ideation scores scored "yes" on items 4 (active suicidal ideation with some intent to act) and/or 5 (active suicidal ideation with specific plan and intent) will be excluded from the study, and if enrolled, will be exited from the study and referred immediately to the nearest emergency mental health facility for additional thorough assessment and appropriate treatment referral.
3. Changes made to treatment regimen within 4 weeks of baseline assessment.
4. Reading level <6th grade as per patient self-report.
5. Patients who have received ECT in the past 2 months prior to Screening.
6. Current pregnancy or breastfeeding
7. Patients must be reasonable medical candidates for ketamine infusion, as determined by a physician co-investigator. Serious, unstable medical illnesses including respiratory [obstructive sleep apnea, or history of difficulty with airway management during previous anesthetics], cardiovascular [including ischemic heart disease and uncontrolled hypertension], and neurologic [including history of severe head injury] will be exclusions.
8. Clinically significant abnormal findings of laboratory parameters [including urine toxicology screen for unreported drugs of abuse], vitals, or ECG.
9. Uncontrolled or poorly controlled hypertension, as determined by a physician co-investigator's review of vitals collected during screening and any other relevant medical history/records.
10. Patients with one or more seizures without a clear and resolved etiology.
11. Patients starting hormonal treatment (e.g., estrogen) in the 3 months prior to Screening.
12. Past intolerance or hypersensitivity to ketamine.
13. Patients taking medications with known activity at the NMDA or AMPA glutamate receptor [riluzole, amantadine, memantine, topiramate, dextromethorphan, D-cycloserine], or the mu-opioid receptor [opiate medications--morphine, oxycodone, heroin, fentanyl)]. However, lamotrigine will not be a study exclusion given that it has been shown not to impact ketamine's safety profile or its antidepressant efficacy.
14. Patients taking any of the following medications: St John's Wort, theophylline, tramadol, metrizamide.
15. Patients who report meditating with mindfulness techniques >1 hour weekly (on average) for the past 6 months or longer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Price, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kheirkhah M, McDonald N, Aepfelbacher J, Rengasamy ML, Shivanekar S, Spotts C, Cooper I, Baumeister A, Bell E, Do-Nguyen K, Woody ML, Hossein S, Henter ID, Nugent AC, Hejazi NS, Jamalabadi H, Yavi M, Walter M, Zarate CA Jr, Price RB. Mindfulness, music, visual occlusion in ketamine therapy for depression: do they change outcomes? A qualitative and quantitative analysis of a randomized controlled trial. Front Psychiatry. 2025 Sep 2;16:1642025. doi: 10.3389/fpsyt.2025.1642025. eCollection 2025. PMID 40964432

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Started | 22 | 21
Completed | 22 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.00 (13.82) | 36.05 (30.29) | 38.07 (13.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 18 | 20 | 38
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 17 | 17 | 34
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Montgomery Asberg Depression Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Clinician-rated depression (range: 0-60; higher scores = worse outcome)
  units on a scale | 30.64 (6.27) | 30.29 (6.21) | 30.47 (6.17)

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale
Description: Clinician-rated depression (range: 0-60; higher scores = worse outcome)
Time Frame: 24hrs post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 20 | 20
score on a scale | 12.50 (7.94) | 13.30 (8.90)

2. Primary Outcome: Montgomery-Asberg Depression Rating Scale
Description: Clinician-rated depression (range: 0-60; higher scores = worse outcome)
Time Frame: 5 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 21 | 20
score on a scale | 15.81 (7.84) | 14.30 (10.69)

3. Primary Outcome: Montgomery-Asberg Depression Rating Scale
Description: Clinician-rated depression (range: 0-60; higher scores = worse outcome)
Time Frame: 12 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 21 | 19
score on a scale | 15.43 (8.42) | 17.21 (11.74)

4. Primary Outcome: Montgomery-Asberg Depression Rating Scale
Description: Clinician-rated depression (range: 0-60; higher scores = worse outcome)
Time Frame: 21 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 19 | 20
score on a scale | 18.90 (11.71) | 17.10 (11.39)

5. Primary Outcome: Montgomery-Asberg Depression Rating Scale
Description: Clinician-rated depression (range: 0-60; higher scores = worse outcome)
Time Frame: 30 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 20 | 20
score on a scale | 18.55 (12.02) | 20.05 (11.64)

6. Primary Outcome: State Mindfulness Scale
Description: Self-reported mindfulness (range 21-105; higher scores = more mindfulness)
Time Frame: 80min post-infusion
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 22 | 21
score on a scale | 77.68 (13.74) | 83.33 (15.27)

7. Secondary Outcome: Modified Hamilton Depression Rating Scale
Description: Clinician-rated depression (range: 0-52; higher scores = worse outcome)
Time Frame: 24hrs post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 20 | 20
score on a scale | 10.00 (5.17) | 9.55 (5.50)

8. Secondary Outcome: Modified Hamilton Depression Rating Scale
Description: Clinician-rated depression (range: 0-52; higher scores = worse outcome)
Time Frame: 5 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 21 | 20
score on a scale | 10.95 (5.13) | 10.15 (6.60)

9. Secondary Outcome: Modified Hamilton Depression Rating Scale
Description: Clinician-rated depression (range: 0-52; higher scores = worse outcome)
Time Frame: 12 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 21 | 19
score on a scale | 10.67 (6.30) | 11.11 (6.32)

10. Secondary Outcome: Modified Hamilton Depression Rating Scale
Description: Clinician-rated depression (range: 0-52; higher scores = worse outcome)
Time Frame: 21 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 19 | 20
score on a scale | 12.05 (7.09) | 11.30 (6.67)

11. Secondary Outcome: Modified Hamilton Depression Rating Scale
Description: Clinician-rated depression (range: 0-52; higher scores = worse outcome)
Time Frame: 30 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 20 | 20
score on a scale | 12.69 (7.42) | 12.45 (6.90)

12. Secondary Outcome: Quick Inventory of Depressive Symptoms
Description: Self-reported depression (range: 0-27; higher scores = worse outcome)
Time Frame: 24hrs post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 20 | 20
score on a scale | 6.55 (5.08) | 6.90 (5.10)

13. Secondary Outcome: Quick Inventory of Depressive Symptoms
Description: Self-reported depression (range: 0-27; higher scores = worse outcome)
Time Frame: 5 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 19 | 19
score on a scale | 8.05 (4.31) | 9.90 (7.58)

14. Secondary Outcome: Quick Inventory of Depressive Symptoms
Description: Self-reported depression (range: 0-27; higher scores = worse outcome)
Time Frame: 12 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 20 | 19
score on a scale | 8.80 (4.94) | 7.95 (5.70)

15. Secondary Outcome: Quick Inventory of Depressive Symptoms
Description: Self-reported depression (range: 0-27; higher scores = worse outcome)
Time Frame: 21 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 19 | 18
score on a scale | 9.68 (5.18) | 8.50 (5.83)

16. Secondary Outcome: Quick Inventory of Depressive Symptoms
Description: Self-reported depression (range: 0-27; higher scores = worse outcome)
Time Frame: 30 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 20 | 17
score on a scale | 9.30 (5.22) | 8.47 (4.94)

17. Secondary Outcome: Hood Mysticism Scale
Description: clinician-administered to assess mystical experiences (range: -64 to +64; higher scores = greater mystical experience)
Time Frame: 40 minutes post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 22 | 21
score on a scale | -.05 (5.59) | .05 (5.70)

18. Secondary Outcome: Mindful Attention Awareness Scale
Description: self-reported trait mindfulness (range: 1-6; higher scores=greater mindfulness)
Time Frame: 24hrs post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 20 | 20
score on a scale | 3.73 (1.05) | 3.80 (.92)

19. Secondary Outcome: Mindful Attention Awareness Scale
Description: self-reported trait mindfulness (range: 1-6; higher scores=greater mindfulness)
Time Frame: 5 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 21 | 19
score on a scale | 3.90 (.80) | 4.15 (.96)

20. Secondary Outcome: Mindful Attention Awareness Scale
Description: self-reported trait mindfulness (range: 1-6; higher scores=greater mindfulness)
Time Frame: 12 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 20 | 19
score on a scale | 3.90 (.92) | 4.09 (.87)

21. Secondary Outcome: Mindful Attention Awareness Scale
Description: self-reported trait mindfulness (range: 1-6; higher scores=greater mindfulness)
Time Frame: 21 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 20 | 18
score on a scale | 3.79 (.73) | 3.86 (1.04)

22. Secondary Outcome: Mindful Attention Awareness Scale
Description: self-reported trait mindfulness (range: 1-6; higher scores=greater mindfulness)
Time Frame: 30 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 20 | 17
score on a scale | 3.81 (.74) | 3.94 (1.04)

23. Secondary Outcome: Daily Spiritual Experience Scale
Description: self-reported spiritual experiences (range: 1-6; higher scores=greater spiritual experience)
Time Frame: 5 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 20 | 19
score on a scale | 2.52 (.95) | 2.20 (.86)

24. Secondary Outcome: Daily Spiritual Experience Scale
Description: self-reported spiritual experiences (range: 1-6; higher scores=greater spiritual experience)
Time Frame: 12 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 20 | 19
score on a scale | 2.51 (1.27) | 2.39 (1.06)

25. Secondary Outcome: Daily Spiritual Experience Scale
Description: self-reported spiritual experiences (range: 1-6; higher scores=greater spiritual experience)
Time Frame: 21 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 20 | 18
score on a scale | 2.36 (1.01) | 2.24 (1.12)

26. Secondary Outcome: Daily Spiritual Experience Scale
Description: self-reported spiritual experiences (range: 1-6; higher scores=greater spiritual experience)
Time Frame: 30 days post-intervention
Population: All participants who were assigned to the arm and were willing and able to complete this specific measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
Number analyzed (Participants) | 20 | 17
score on a scale | 2.52 (1.17) | 2.34 (.98)

27. Other Pre Specified Outcome: Sustained Attention Response Task (SART) Omission Errors
Description: performance-based measure of mindful attention
Time Frame: infusion +24 hours (1 day)
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Sustained Attention Response Task (SART) Self-reported Task Focus
Description: self-report rating of being on-task (range: 1-7; higher score=more on-task)
Time Frame: infusion +24 hours (1 day)
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Awe Experience Scale
Description: self-report measure of awe-inspiring experiences (range: 30-210; higher score=greater awe)
Time Frame: infusion +80min
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Dual Probe Video Task
Description: attentional bias (proportion score) towards sad film clips (range: 0-1.0; higher score=greater attention bias towards sad films)
Time Frame: infusion +24 hours (1 day)
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Pain Rating Via Quantitative Sensory Testing
Description: Pain rating obtained from Quantitative Sensory Testing by mechanical temporal summation (range: 0-10; higher score=more pain)
Time Frame: 1-hour post-infusion
Reporting Status: Not Posted

32. Other Pre Specified Outcome: PROMIS Pain Intensity Score
Description: PROMIS Pain Intensity Short Form scale T-score (range=0-100; higher score=worse pain)
Time Frame: 1-hour post-infusion
Reporting Status: Not Posted

33. Other Pre Specified Outcome: PROMIS Pain Interference Score
Description: PROMIS Pain Interference Short Form scale T-score (range=0-100; higher score=worse pain)
Time Frame: 1-hour post-infusion
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 hours
Description: Adverse events were collected using the Patient Rated Inventory of Side Effects (PRISE; Rush et al 2004) instrument and the Clinician-Administered Dissociative States Scale (CADSS). Open-ended questions were also used to inquire about any additional adverse events not captured on the PRISE. Adverse events were tallied for all symptoms that were reported as new or worsening from pre-infusion baseline with onset during the infusion and/or within the subsequent 24hr period.
Arm/Group | Intravenous Ketamine + Mindfulness Exercises | Intravenous Ketamine + Academic Exercises
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 22/22 | 21/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous Ketamine + Mindfulness Exercises (N=22) | Intravenous Ketamine + Academic Exercises (N=21)
anxiety (Psychiatric disorders) | 2 | 1
decreased energy (General disorders) | 3 | 7
diarrhea (Gastrointestinal disorders) | 6 | 1
difficulty sleeping: too little (Psychiatric disorders) | 4 | 2
difficulty sleeping: too much (Psychiatric disorders) | 2 | 1
dissociative symptoms (Psychiatric disorders) | 20 | 21
dizziness (Nervous system disorders) | 9 | 14
dry mouth (Gastrointestinal disorders) | 7 | 9
elevated blood pressure (Vascular disorders) | 1 | 0
emotional indifference (Psychiatric disorders) | 3 | 1
headache (Nervous system disorders) | 4 | 5
increased appetite (Gastrointestinal disorders) | 10 | 7
increased weight (Metabolism and nutrition disorders) | 3 | 0
loss of sexual desire (Reproductive system and breast disorders) | 3 | 0
nausea (Gastrointestinal disorders) | 4 | 6
palpitations (Cardiac disorders) | 4 | 2
restlessness (General disorders) | 5 | 3
sweating (General disorders) | 5 | 1
tremors (Nervous system disorders) | 1 | 1
trouble achieving orgasm (Reproductive system and breast disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
Pilot study leading to small numbers of patients in each treatment arm. Descriptive statistics are reported without statistical analysis to directly compare groups, given the small number of patients within each group leading to low statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT05168735/Prot_SAP_000.pdf